CLINICAL TRIAL: NCT06170437
Title: Healthy Homes Study: A Protocol for a Place-based Smoke-free Home Intervention in Federally Subsidized Housing
Brief Title: Smoke-free Home Study in Subsidized Housing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24631; R01MD016898 (NIH)
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Tobacco Dependence; Tobacco Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The study's investigators will train bilingual study staff to deliver the intervention to residents using a script that matches the content in the smoke-free home intervention pamphlet. The in-person delivery of the intervention and pamphlet will be the primary modes of intervention delivery to residents. The pamphlet will include: (1) the harms of tobacco, e-cigarette use, cannabis use and exposure (secondhand and thirdhand), (2) an exercise to calculate personal cost of tobacco use, (3) benefits of a smoke-free home, (4) skill-building on how to adopt a smoke-free home, and (5) motivational language on smoke-free home adoption. The study staff will qualitatively assess participants' knowledge by prompting questions on the topics covered and will refer participants to lay-health workers (LHWs) for one-on-one coaching. Participants will receive a pledge to designate their homes smoke-free.
  Interventions: Behavioral: Smoke-free home resident intervention; Behavioral: Lay Health Worker coaching
- Waitlist Control Group (No Intervention): The current standard of care does not include any interventions for smoke-free home adoption or referrals to tobacco treatment resources. At the end of the primary endpoint (6 months), control participants will be offered the intervention.

INTERVENTIONS:
Behavioral: Smoke-free home resident intervention — Study staff delivered intervention on how to adopt a smoke free home using a pamphlet
  Arms: Intervention
Behavioral: Lay Health Worker coaching — Brief tobacco cessation coaching by lay health worker housing staff with residents within 2 weeks of the smoke-free home resident intervention, and on a monthly schedule as part of their routine encounters with residents (total 6 sessions).
  Arms: Intervention

SUMMARY:
Comprehensive smoke-free policies have the potential to substantially reduce tobacco-related disparities among populations in subsidized housing. This study fills this gap by identifying approaches to increase the implementation of smoke-free policies in all types of subsidized housing by increasing the voluntary adoption of smoke-free homes and promoting access to smoking cessation services.

DETAILED DESCRIPTION:
OBJECTIVES:

The investigators will build on previous studies, where a smoke-free home intervention to increase voluntary adoption of smoke-free homes in permanent supportive housing for formerly homeless adults was developed and evaluated.

Aim 1: To estimate the effect of our adapted smoke-free home intervention on the primary outcome of residents' voluntary adoption of smoke-free homes and the secondary outcome of biochemically-verified tobacco abstinence at 6-months follow-up.

Aim 2: To determine the cost of our adapted smoke-free home intervention and determine whether it is a cost-effective use of health care resources.

Aim 3: To evaluate variation in stakeholders' perspectives on the adapted smoke-free home intervention's adaptability, scalability and sustainability.The proposed intervention can expand access to smoke-free policies and smoking cessation services in subsidized housing, thereby reducing racial/ethnic disparities in tobacco use, tobacco exposure and chronic disease in these populations.

OUTLINE:

A wait-list cluster randomized controlled trial of the adapted smoke-free home intervention compared to usual care among residents from subsidized housing sites in Northern California. Participants from twenty-four subsidized housing sites will be randomized into intervention and waitlist control arms

ELIGIBILITY:
Inclusion Criteria:

Eligible resident participants

* Current smokers defined as:

  * Smoked at least 100 cigarettes in lifetime
  * Smoked daily in the past 7 days, and at least 5 cigarettes per day, verified by expired CO ≥ 5 parts per million [ppm] Smokerlyzer CO+ monitor),
  * Smoke in their home
* Expect to live in the subsidized housing site for at least 12 months
* Age ≥ 18 years
* Speak Chinese (Cantonese or Mandarin), English, Spanish, or Vietnamese
* Able to provide informed consent.

Exclusion Criteria:

* Contraindication to any study-related procedures or assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 544 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants adopting a smoke-free home for ≥90 days | 6 months
  The percentage of participants who reported to adopt a smoke-free home in the past 90 days will be reported

SECONDARY OUTCOMES:
Percentage of participants with point prevalent abstinence (PPA) | 6 months
  The percentage of participants with carbon dioxide (CO)-verified tobacco abstinence will be reported at the 6 month follow-up visit.

OTHER OUTCOMES:
Percentage of participants adopting a cannabis-free home among cannabis users | 6 months
  The percentage of participants who reported to adopt a cannabis-free home in the past 90 days will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Maya Vijayaraghavan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets may be provided to other researchers upon request and approval by the investigator

REFERENCES:
- [Derived] Hawes MR, Chakravarty D, Cheng J, Handley MA, Tsoh JY, Lin TK, Hiatt RA, Vijayaraghavan M. The Healthy Homes Study: Protocol for a cluster randomized trial of a place-based smoke-free home intervention in affordable housing. PLoS One. 2025 Jul 29;20(7):e0328786. doi: 10.1371/journal.pone.0328786. eCollection 2025. PMID 40729126